CLINICAL TRIAL: NCT01854528
Title: A Randomized, Open-Labeled Study to Evaluate the Efficacy and Safety of ABT-450/Ritonavir/ABT-267 and ABT-333 Co-administered With Ribavirin Compared to Telaprevir Co-administered With Pegylated Interferon a-2a and Ribavirin in Treatment-Experienced Adults With Chronic Hepatitis C Genotype 1 Virus Infection (MALACHITE-II)
Brief Title: A Study to Evaluate the Efficacy and Safety of Three Experimental Drugs Compared With Telaprevir (a Licensed Product) for Treatment of Chronic Hepatitis C Infection in Treatment-experienced Adults
Acronym: MALACHITE II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M13-862; 2012-003738-18 (EudraCT Number)
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2016-06

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Partial responder; Interferon free; Treatment-experienced; Relapser; Hepatitis C Virus; Null responder; Hepatitis C Genotype 1; paritaprevir; ombitasvir; dasabuvir; ribavirin; Viekira PAK; Chronic hepatitis C
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — dasabuvir; ombitasvir; paritaprevir; Viekira Pak; Ribavirin; telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3-DAA/RBV (Experimental): 3-DAA (ABT-450/r/ABT-267 [150 mg/ 100 mg/ 25 mg once daily] and ABT-333 [250 mg twice daily]) plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks.
  Interventions: Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin
- TPV/RBV (Active Comparator): TPV (750 mg every 8 hours) coadministered with pegIFN (180 micrograms subcutaneously [SC] weekly) and weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks, followed by pegIFN (180 micrograms SC weekly) and weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for either 12 or 36 weeks, per local prescribing information.
  Interventions: Drug: Ribavirin; Drug: Pegylated Interferon a-2a (PegINF); Drug: Telaprevir

INTERVENTIONS:
Drug: ABT-450/r/ABT-267, ABT-333 — Tablet; ABT-450 coformulated with ritonavir and ABT-267, ABT-333 tablet
  Other Names: ABT-267 also known as ombitasvir; ABT-450 also known as paritaprevir; ABT-333 also known as dasabuvir; Viekira PAK
  Arms: 3-DAA/RBV
Drug: Ribavirin — Tablet
Drug: Pegylated Interferon a-2a (PegINF) — Pre-filled syringe
  Arms: TPV/RBV
Drug: Telaprevir — Film-coated tablet
  Arms: TPV/RBV

SUMMARY:
The purpose of this study is to evaluate the safety and antiviral activity of 3 direct-acting antiviral agents (DAAs; ABT-450/ritonavir/ABT-267 [ABT-450/r/ABT-267; ABT-267 also known as ombitasvir] and ABT-333 [also known as dasabuvir]) plus ribavirin (RBV) compared with telaprevir (TPV) with pegylated interferon/ribavirin (pegIFN/RBV) in patients with chronic hepatitis C virus genotype 1 (HCV GT1) infection without cirrhosis who were previously treated with pegylated interferon/ribavirin (pegIFN/RBV).

DETAILED DESCRIPTION:
A randomized, open-label, parallel-arm, multicenter study to evaluate the safety and antiviral activity of the 3-DAA regimen (ABT-450/ritonavir/ABT-267 [ABT-450/r/ABT-267] and ABT-333) plus ribavirin (3-DAA/RBV) compared with the combination of telaprevir (TPV) with RBV and pegIFN (TPV/RBV) in noncirrhotic participants with chronic hepatitis C virus genotype 1 (HCV GT1) infection who were previously treated with pegylated interferon/ribavirin (pegIFN/RBV).

Participants were randomized in a 2:1 ratio to receive 3-DAA/RBV (ABT-450/r/ABT-267 and ABT-333 plus RBV for 12 weeks) or TPV/RBV (TPV co-administered with pegIFN and RBV for 12 weeks, followed by followed by pegIFN and RBV for either 12 or 36 weeks, per local prescribing information).

ELIGIBILITY:
Inclusion Criteria:

* Females must be practicing specific forms of birth control on study treatment, or be post-menopausal for more than 2 years or surgically sterile
* Chronic hepatitis C infection (positive for anti-HCV antibody or HCV RNA at least 6 months before screening and at the time of screening; or positive for anti-HCV antibody or HCV RNA at the time of screening with a liver biopsy consistent with chronic HCV infection)
* Screening laboratory result indicating HCV genotype 1 infection (HCV GT1)
* Participant must have documentation of adherence to a prior pegIFN/RBV combination therapy and meet one of the protocol definitions for treatment failure: null responder, partial responder, relapser
* No evidence of liver cirrhosis

Exclusion Criteria:

* Positive hepatitis B surface antigen or anti-human immunodeficiency virus antibody
* Positive screen for drugs or alcohol
* Significant sensitivity to any drug
* Use of contraindicated medications within 2 weeks of dosing
* Abnormal laboratory tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Luo, MD, Study Director — AbbVie

REFERENCES:
- [Result] Dore GJ, Conway B, Luo Y, Janczewska E, Knysz B, Liu Y, Streinu-Cercel A, Caruntu FA, Curescu M, Skoien R, Ghesquiere W, Mazur W, Soza A, Fuster F, Greenbloom S, Motoc A, Arama V, Shaw D, Tornai I, Sasadeusz J, Dalgard O, Sullivan D, Liu X, Kapoor M, Campbell A, Podsadecki T. Efficacy and safety of ombitasvir/paritaprevir/r and dasabuvir compared to IFN-containing regimens in genotype 1 HCV patients: The MALACHITE-I/II trials. J Hepatol. 2016 Jan;64(1):19-28. doi: 10.1016/j.jhep.2015.08.015. Epub 2015 Aug 29. PMID 26321288
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 154 participants were randomized: 6 participants did not receive at least 1 dose of study drug and were excluded from the analyses; 148 participants received at least 1 dose and were included in the intent-to-treat (ITT) population.
Period: Overall Study
Arm/Group | 3-DAA/RBV | TPV/RBV
Started | 101 | 47
Completed | 101 | 32
Not Completed | 0 | 15
Not completed — Adverse Event | 0 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Virologic Failure | 0 | 9

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug (ITT population) were included in baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | 3-DAA/RBV | TPV/RBV | Total
Number analyzed (Participants) | 101 | 47 | 148
Age, Continuous [Median (Standard Deviation); unit: years] | 46.9 (12.15) | 45.0 (10.35) | 46.3 (11.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 19 | 65
  Male | 55 | 28 | 83

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Treatment
Description: The percentage of participants with sustained virologic response (plasma Hepatitis C virus ribonucleic acid [HCV RNA] level less than the lower limit of quantitation [< LLOQ]) 12 weeks after the last dose of study drug. The LLOQ for the assay was 25 IU/mL.
Time Frame: 12 weeks after the last dose of study drug
Population: ITT population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 3-DAA/RBV | TPV/RBV
Number analyzed (Participants) | 101 | 47
percentage of participants | 100.0 | 66.0
Statistical Analysis 1: Comparison: 3-DAA/RBV vs TPV/RBV; P-value for the difference in sustained virologic response rates 12 weeks after the last dose between treatment groups with HCV subgenotype (1a, non-1a) from stratum adjusted Mantel-Haenszel with previous type of response to pegIFN/RBV treatment (relapser, partial or null responder) as strata; Test type: Superiority or Other; p < 0.001, Stratum adjusted Mantel-Haenszel; Mean Difference (Final Values) = 34.26, 95% CI 2-sided [21.09 to 47.42]

2. Secondary Outcome: Mean Change From Baseline to Final Treatment Visit in the Mental Component Summary (MCS) Score of the Short-Form 36 Health Survey - Version 2 (SF-36v2)
Description: The SF-36v2 is a general health-related quality of life (HRQoL) instrument with extensive use in multiple disease states. The SF-36v2 instrument comprises a total of 36 items (questions) targeting a participant's functional health and well-being in 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health). Domain scores were aggregated into an MCS score (from 0 to 100; a higher score indicates better mental function and well-being).
Time Frame: Baseline and Final Treatment Visit (up to Week 12 for 3-DAA/RBV and up to Week 24 or 48 for TPV/RBV)
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 3-DAA/RBV | TPV/RBV
Number analyzed (Participants) | 101 | 45
units on a scale | -1.3 (8.32) | -9.8 (11.05)
Statistical Analysis 1: Comparison: 3-DAA/RBV vs TPV/RBV; P-value from ANCOVA model including baseline score and region as covariates and treatment arm as a factor; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 8.64, 95% CI 2-sided [5.43 to 11.85]

3. Secondary Outcome: Mean Change From Baseline to Final Treatment Visit in the Physical Component Summary (PCS) Score of the Short-Form 36 Health Survey - Version 2 (SF-36v2)
Description: The SF-36v2 is a general health-related quality of life (HRQoL) instrument with extensive use in multiple disease states. The SF-36v2 instrument comprises a total of 36 items (questions) targeting a participant's functional health and well-being in 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health). Domain scores were aggregated into a PCS score (range = 0 to 100; a higher score indicates better mental function and well-being).
Time Frame: Baseline and Final Treatment Visit (up to Week 12 for 3-DAA/RBV and up to Week 24 or 48 for TPV/RBV)
Population: All participants in the ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 3-DAA/RBV | TPV/RBV
Number analyzed (Participants) | 101 | 45
units on a scale | 0.4 (7.16) | -7.7 (7.72)
Statistical Analysis 1: Comparison: 3-DAA/RBV vs TPV/RBV; P-value from ANCOVA model including baseline score and region as covariates and treatment arm as a factor; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = 7.55, 95% CI 2-sided [5.11 to 9.98]

4. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks After Treatment
Description: The percentage of participants with sustained virologic response (plasma Hepatitis C virus ribonucleic acid [HCV RNA] level less than the lower limit of quantitation [< LLOQ]) 24 weeks after the last dose of study drug. The LLOQ for the assay was 25 IU/mL.
Time Frame: 24 weeks after the last dose of study drug
Population: All participants in the ITT population with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | 3-DAA/RBV | TPV/RBV
Number analyzed (Participants) | 101 | 47
percentage of participants | 99.0 | 66.0
Statistical Analysis 1: Comparison: 3-DAA/RBV vs TPV/RBV; P-value from logistic regression model including treatment arm, baseline log10 HCV RNA level, HCV subgenotype, and previous response to pegIFN/RBV treatment as predictors; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 54.7, 95% CI 2-sided [6.9 to 435.1]

5. Secondary Outcome: Percentage of Participants With Virologic Failure During Treatment
Description: Virologic failure during treatment was defined as HCV ribonucleic acid (RNA) confirmed greater than or equal to the lower limit of quantification (≥ LLOQ) after HCV RNA < LLOQ during treatment or confirmed HCV RNA ≥ LLOQ at the end of treatment.
Time Frame: Baseline to end of treatment (12 weeks for 3-DAA/RBV and 24 or 48 weeks for TPV/RBV)
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3-DAA/RBV | TPV/RBV
Number analyzed (Participants) | 101 | 47
percentage of participants | 0 [0.0 to 3.7] | 19.1 [7.9 to 30.4]

6. Secondary Outcome: Percentage of Participants With Virologic Relapse After Treatment
Description: Participants who completed treatment with plasma HCV RNA less than the lower limit of quantification (<LLOQ) at the end of treatment were considered to have virologic relapse if they had confirmed HCV RNA ≥ LLOQ during the post-treatment period.
Time Frame: Between end of treatment (Week 12 for 3-DAA/RBV and Week 24 or 48 for TPV/RBV) and Post-treatment (up to Week 12 Post-treatment)
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3-DAA/RBV | TPV/RBV
Number analyzed (Participants) | 101 | 47
percentage of participants | 0 [0.0 to 3.7] | 6.3 [0.0 to 14.6]

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of study drug administration to 30 days after last dose of study drug (up to 52 weeks); SAEs were also collected from the time that informed consent was obtained until the end of the study (total up to 101 weeks).
Description: AEs were collected from first dose to 30 days after last dose (16 weeks for 12-week treatment, 28 weeks for 24-week treatment, 52 weeks for 48-week treatment); SAEs were collected from the time that informed consent was obtained to end of study (up to 65 weeks for 12-week treatment, 77 weeks for 24-week treatment, 101 weeks for 48-week treatment).
Arm/Group | 3-DAA/RBV | TPV/RBV
Serious Adverse Events (participants affected / at risk) | 1/101 | 5/47
Other Adverse Events (participants affected / at risk) | 54/101 | 43/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3-DAA/RBV (N=101) | TPV/RBV (N=47)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
INJECTION SITE PHLEBITIS (General disorders) | 0 | 1
APPENDICITIS (Infections and infestations) | 1 | 0
DIARRHOEA INFECTIOUS (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 | 1
EPILEPSY (Nervous system disorders) | 1 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3-DAA/RBV (N=101) | TPV/RBV (N=47)
ANAEMIA (Blood and lymphatic system disorders) | 3 | 14
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 5
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 12
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 4
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 4
ANAL PRURITUS (Gastrointestinal disorders) | 0 | 12
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 | 3
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 3
NAUSEA (Gastrointestinal disorders) | 10 | 20
VOMITING (Gastrointestinal disorders) | 3 | 7
ASTHENIA (General disorders) | 8 | 16
CHEST PAIN (General disorders) | 0 | 3
CHILLS (General disorders) | 3 | 5
FATIGUE (General disorders) | 12 | 12
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 3
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 4
INJECTION SITE ERYTHEMA (General disorders) | 0 | 3
PYREXIA (General disorders) | 2 | 15
GASTROENTERITIS (Infections and infestations) | 2 | 3
NASOPHARYNGITIS (Infections and infestations) | 5 | 5
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 | 8
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 8
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 9
DIZZINESS (Nervous system disorders) | 5 | 7
DYSGEUSIA (Nervous system disorders) | 1 | 4
HEADACHE (Nervous system disorders) | 29 | 21
LETHARGY (Nervous system disorders) | 5 | 3
PARAESTHESIA (Nervous system disorders) | 0 | 3
DEPRESSED MOOD (Psychiatric disorders) | 0 | 3
DEPRESSION (Psychiatric disorders) | 0 | 3
INSOMNIA (Psychiatric disorders) | 6 | 10
IRRITABILITY (Psychiatric disorders) | 2 | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 | 12
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 3
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 6
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 7
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 3
PRURITUS (Skin and subcutaneous tissue disorders) | 13 | 19
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 3
RASH (Skin and subcutaneous tissue disorders) | 3 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.